CLINICAL TRIAL: NCT02143024
Title: A Family-based Primary Care Intervention to Enhance Older Men's Depression Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of Washington (Other); RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 807849
Record Dates: First submitted 2013-06-19; First posted 2014-05-20 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Major Depression
Keywords: depression; family; primary health care
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-based depression intervention (Experimental): The family-focused component will consist of up to up to 10 joint (i.e. older man alone and/or with family members) sessions that will cover specific topics related to family support of men's depression care provided by a clinic-based social worker
  Interventions: Behavioral: Family-based depression intervention
- Usual care plus educational materials (Active Comparator): Control subjects will receive usual care in the clinic enhanced by a single depression psychoeducation session.
  Interventions: Behavioral: Usual care plus educational materials

INTERVENTIONS:
Behavioral: Family-based depression intervention — The primary focus of our approach is on effectively engaging family members of depressed older men in the care of the patient. The interventionist (social worker) will 1) work jointly with a family member and older men to strengthen depression self-management and participation during primary care visits and 2) conduct a brief training module for primary care provider skills to strengthen their skills in working with family members.
  Arms: Family-based depression intervention
Behavioral: Usual care plus educational materials — Control subjects will receive usual care in the clinic augmented by psychoeducation. Family members will be given standard psychoeducational materials on depression.
  Arms: Usual care plus educational materials

SUMMARY:
Despite the public health importance of clinical depression, more than 50% of depressed adults receive inadequate or no treatment, with even higher rates of under-treatment in men and minorities. Family members and/or friends often assist older adults in their health care and may help overcome barriers to formal care, yet there is a lack of primary care-based interventions that mobilize family members and friends to improve depression treatment. In partnership with a community-based clinic, this research will address this scientific gap by developing and then testing the feasibility and acceptability of a family-based intervention that can be delivered pragmatically in a primary care setting serving large numbers of older minorities.

DETAILED DESCRIPTION:
The family-based intervention will be tested in a 6 month randomized controlled trial of 24 depressed older men-family member dyads (18 intervention and 6 controls). The purpose of the RCT is to test the acceptability of the intervention, as well as the feasibility of the study methods. Patients from the RCT will be identified from a family practice clinic based on their scores on the PHQ-9 as well as additional inclusion and exclusion criteria. Once they and their family member have agreed to participate, patients will be randomized either to the family based intervention or a usual care control condition augmented by family psychoeducation. The investigators will recruit English and Spanish speaking age 60 and above older men from SJGH who have 1) significant depressive symptoms (i.e. PHQ > 15, 2) have at least one criteria A symptom (depressed mood or anhedonia), 3) depression-related functional impairment) and 4) an adult family member willing to participate in the study. We have chosen a higher cut-off to minimize false positives. We will exclude psychotic, demented or institutionalized men. After enrollment, 24 dyads (i.e. older man and family member) will be randomized one of two groups: intervention or usual care augmented by written psychoeducational materials on depression. Dyads will be randomized to achieve a 2:1 ratio of intervention versus usual care dyads (i.e. 18 intervention and 6 control dyads). To ensure adequate numbers of ethnic minority patients in each arm of the trial, we will conduct a stratified randomization such that each arm of the RCT is 50% English language preferring and 50% Spanish language preferring (i.e. 3 in control and 9 in intervention arm). The research assistant will conduct subject assessment at baseline, 1-month, 3-months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Men, age 50 and above
* English or Spanish speaking
* Score of >9 on the PHQ-9
* Non-demented
* Have an adult family member or close friend who can participate

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ladson Hinton, MD, Principal Investigator — University of California, Davis
Locations (1):
- San Joaquin General Hospital, Stockton, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 people were referred to the study. 41 people were assessed, 4 were not assessed for eligibility. 18 were excluded; 10 did not meet inclusion criteria and 8 declined. A total of 23 people were randomized as part of the study.
Period: Overall Study
Arm/Group | Family-based Depression Intervention | Usual Care Plus Educational Materials
Started | 15 | 8
Received Treatment (These people were randomized and received at least 1 session before dropping out of the study.) | 13 | 7
Completed | 13 | 7
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants that received at least 1 session.
Groups:
- Total: Total of all reporting groups
Arm/Group | Family-based Depression Intervention | Usual Care Plus Educational Materials | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (9.6) | 57.4 (4.8) | 59.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 7 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 10 | 2 | 12
  African American | 1 | 3 | 4
  White | 1 | 1 | 2
  Native American and White | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms
Description: Patient Health Questionnaire (PHQ-9) scale; 0-27 scoring units; higher scores indicate more severe depressive symptoms.
Time Frame: baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Family-based Depression Intervention | Usual Care Plus Educational Materials
Number analyzed (Participants) | 13 | 7
units on a scale
  baseline | 14.8 (2.9) | 15.3 (4.1)
  3 months | 10.1 (6.6) | 13.0 (7.5)
  6 months | 11.8 (7.1) | 13.3 (6.3)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored up until the 6 month visit.
Arm/Group | Family-based Depression Intervention | Usual Care Plus Educational Materials
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes